CLINICAL TRIAL: NCT06060743
Title: Examining the Effect of the Mobile Application Developed for Individuals With Type 2 Diabetes Using Insulin on the Perception of Insulin Use and Self-Management
Brief Title: Examining the Effect of Mobile Application on Insulin Use Perception and Self-Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Nedime Hazal Döner, lecturer, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: EU-NF-NHD-01
Record Dates: First submitted 2023-09-25; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Type 2 Diabetes Treated With Insulin
Keywords: type 2 diabetes mellitus; mobile application; Self-Management
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: It consists of two groups, application and control, and three follow-ups.
Who Masked: Participant, Outcomes Assessor
Masking Description: In the study, groups were determined by block randomization. The randomization list was created by block randomization according to age and gender.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Data collection tools were applied to individuals in the control group on day 0 (Z0), day 14 (Z1) and day 28 (Z2) of follow-up. Data collection tools applied to the control group are as follows: Patient Introduction Form, Insulin Treatment Appraisal Scale,, Insulin Therapy Self-Management Scale, Insulin Information Form, Insulin Injection Skill Observation Form and Metabolic Control Variables Form.
- application group (Experimental): Individuals in the application group will be given individual training on how to use the application through the application demo. Data collection forms will be applied to individuals in the application group on day 0 (Z0), day 14 (Z1) and day 28 (Z2). The forms to be used are: Patient Introduction Form, Insulin Treatment Appraisal Scale, Insulin Therapy Self-Management Scale, Insulin Information Form, Metabolic Control Variables Form, Insulin Injection Skill Observation Form and Digital Literacy Scale.
  Interventions: Other: INS-MOBILE: Mobile Application Developed for Insulin Use

INTERVENTIONS:
Other: INS-MOBILE: Mobile Application Developed for Insulin Use — After determining the application and control groups in the research, the purpose of the research was explained to both groups. Participants were informed that the application would last 1 month. It was explained that data collection forms would be filled out before the application (Z0), on the 14th day of the application (Z1), and on the 28th day of the application (Z2). On the 0th and 28th days of the follow-up, the participants' insulin administration skills were evaluated face-to-face by the researcher using the Insulin Therapy Skill Observation Form. In addition to the standard training given by diabetes training nurses, a mobile application on insulin use was sent to the application group, while the control group was given standard training only by diabetes training nurses.
  Arms: application group

SUMMARY:
The main purpose of the research is; To develop a mobile application for individuals with Type 2 diabetes who use insulin and to examine the effect of the developed mobile application on the perception and self-management of insulin use.

DETAILED DESCRIPTION:
In recent years, an increase in insulin use has been observed in individuals with Type 2 DM. Since any mistake in insulin use can lead to hyperglycemic crisis or severe hypoglycemia, correct administration of insulin forms the basis of successful diabetes management. Errors related to insulin therapy are defined as important and correctable medication errors. Such errors related to insulin therapy can potentially occur at every step of diabetes management.

It is stated that interventions that can provide effective self-management and behavioral change can be planned by evaluating individuals' perceptions of the disease and treatment in diabetes management. In our country, only one thesis study evaluating the effect of video-supported teaching given to type 2 diabetic patients on insulin self-management and application skills has been found. This study found that video-assisted instruction given to patients with Type 2 diabetes increased their ability to administer insulin injections and their self-management. In the thesis study in question, the video was shot by the researcher using a model, and individuals who had been using insulin for at least one year were included in the study. In this project, a mobile application for insulin use will be developed and this application will include three separate videos, two of which are animation videos, and a game for insulin use. Our study will be conducted on individuals who will use insulin for the first time, and no study has been found in our country with this sample and population.

When global goals for sustainable development are examined, it is aimed to "promote mental health and well-being by reducing premature deaths from non-communicable diseases by one third through prevention and treatment by 2030". The development of technology and its availability in every aspect of life has also affected patient care, and technological devices and mobile applications have been integrated into patient care. Studies show that the mobile applications used are effective in managing the disease and maintaining self-care activities in individuals with Type 2 DM. In chronic disease management, both compliance with treatment and self-management can be made permanent with mobile applications developed specifically for the disease.

In the research, the educational material was created with an animated video, and the created video was transferred to the mobile application. Thus, the patient will be able to access the educational content via the mobile application at any time and experience the insulin administration steps countless times on the mobile application. By giving feedback from the application regarding the mistakes made during the application, the user will be able to see at what point he made a mistake. Audiovisual materials used in patient education positively affect learning because they appeal to more than one sensory organ. Utilizing technology and using visual and auditory stimuli in patient education will strengthen learning, and the skills aimed to be acquired with the educational material will become more permanent.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* Aware and communicative,
* Those diagnosed with Type 2 DM and using insulin for the first time
* Able to administer insulin on his own,
* Able to use Android based phone,
* Having a digital literacy scale score above 17,
* Agreeing to participate in the research

Exclusion Criteria:

* Under 18 years of age,
* Having vision problems,
* Do not have an Android phone,
* Unconscious and unable to communicate,
* Not having sufficient motor skills,
* Those who did not agree to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
insulin information sheet | two weeks
  This form, created by the researchers after literature review, consists of 25 questions. This form includes questions about general information about insulins, insulin storage conditions, injection preparation stages, injection sites and injection technique. The form is answered as True/False. The questions in the form were evaluated out of 100 points.

SECONDARY OUTCOMES:
Insulin Treatment Appraisal Scale | two weeks
  The scale consists of two subscales, positive and negative attitude, and 20 items. Scale items are rated on a Likert type scale between "strongly disagree", 1 point, and "strongly agree", 5 points.
Insulin Therapy Self-Management Scale | two weeks
  The scale consists of 32 items with a three-factor structure, scored using a five-point Likert-type scale.
Insulin Injection Skill Observation Form | Evaluated at first and last follow-up/ four weeks
  It consists of 21 items including the stages of insulin injection.

CONTACTS AND LOCATIONS:
Overall Officials: Nedime Hazal Doner, Principal Investigator — Ege University
Locations (1):
- Ege University, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No